CLINICAL TRIAL: NCT02460159
Title: A Phase III, Clinical Trial to Assess the Long Term Safety and Tolerability of MK-0653C in Japanese Patients With Hypercholesterolemia Who Have Inadequate LDL-C Control on Ezetimibe or Atorvastatin Calcium Monotherapy
Brief Title: A Clinical Trial to Assess the Long Term Safety and Tolerability of MK-0653C in Japanese Participants With Hypercholesterolemia (MK-0653C-384)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0653C-384; 152982 (Registry Identifier: JAPIC)
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Results first posted 2018-01-11 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Heterozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EZ 10 mg/Atorva 10 mg FDC (Experimental): one EZ 10 mg/Atorva 10 mg fixed-dose combination (FDC) tablet orally with food once daily for 52 weeks.
  Interventions: Drug: EZ 10 mg/Atorva 10 mg FDC
- EZ 10 mg/Atorva 20 mg FDC (Experimental): one EZ 10 mg/Atorva 20 mg fixed -dose combination (FDC) tablet orally with food once daily for 52 weeks.
  Interventions: Drug: EZ 10 mg/Atorva 20 mg FDC

INTERVENTIONS:
Drug: EZ 10 mg/Atorva 20 mg FDC
  Other Names: MK-0653C
  Arms: EZ 10 mg/Atorva 20 mg FDC
Drug: EZ 10 mg/Atorva 10 mg FDC
  Other Names: MK-0653C
  Arms: EZ 10 mg/Atorva 10 mg FDC

SUMMARY:
This study will assess the safety and tolerability of Ezetimibe (EZ) 10 mg/Atorvastatin (Atora) 10 mg and EZ 10mg/Atora 20 mg fixed-dose combination (FDC) in Japanese participants with hypercholesterolemia uncontrolled with monotherapy of Ezetimibe 10 mg or Atorvastatin up to 20 mg. There is no formal hypothesis for the study.

ELIGIBILITY:
Inclusion Criteria

* Japanese
* Outpatient with hypercholesterolemia
* Has familial hypercholesterolemia (FH) diagnosed per genetic testing or meets two or more of the below criteria based on Japan Atherosclerosis Society Guideline 2012 (JAS2012): Hyper low-density lipoprotein (LDL)-cholesterolemia (an untreated LDL-C level of ≥180mg/dL); tendon xanthoma (tendon xanthoma on the backs of the hands, elbows, knees, etc. or achilles tendon hypertrophy) or xanthoma tuberosum; family history of FH or premature coronary arterial disease (within the participant's second degree relatives)
* Females must be of non-reproductive potential or agree to remain abstinent or use (or partner use) two acceptable methods of birth control from date of signed informed consent to the 14 days after the last dose of study drug
* Agree to maintain a stable diet that is consistent with the JAS 2012 for prevention of atherosclerotic cardiovascular diseases for the duration of the study

Exclusion Criteria

* Uncontrolled hypertension
* Type 1 or uncontrolled type 2 diabetes mellitus (treated or untreated)
* Homozygous familial hypercholesterolemia or has undergone LDL apheresis
* Had a gastrointestinal tract bypass, or other significant intestinal malabsorption
* History of cancer within the past 5 years except for successfully treated dermatological basal cell or squamous cell carcinoma or in situ cervical cancer
* Human immunodeficiency virus (HIV) positive
* History of drug/ alcohol abuse within the past 5 years or psychiatric illness not adequately controlled and stable on pharmacotherapy
* Consumes more than 25 g of alcohol per day
* Consumes more than 1L of grapefruit juice per day
* Currently following an excessive weight reduction diet
* Engaging in a vigorous exercise regimen (e.g.; marathon training, body building training etc.) or intends to start training during the study
* Hypersensitivity or intolerance to ezetimibe or atorvastatin
* History of myopathy or rhabdomyolysis with ezetimibe or any statin
* Pregnant or lactating
* Taking any other investigational drugs and/or has taken any investigational drugs within 30 days

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Teramoto T, Yokote K, Nishida C, Tershakovec A, Oshima N, Takase T, Hirano T. A Phase III open-label clinical trial to assess the long-term safety of ezetimibe and atorvastatin combination therapy in Japanese patients with hypercholesterolemia. J Clin Therapeut Med. 2017;33(8):655-670.

RESULTS

PARTICIPANT FLOW:
Groups:
- EZ 10 mg/Atorva 10 mg FDC: One ezetimibe (EZ) 10 mg/atorvastatin (Atorva) 10 mg fixed-dose combination (FDC) tablet orally with food once daily for 52 weeks.
Period: Overall Study
Arm/Group | EZ 10 mg/Atorva 10 mg FDC | EZ 10 mg/Atorva 20 mg FDC
Started | 117 | 18
Completed | 111 | 17
Not Completed | 6 | 1
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EZ 10 mg/Atorva 10 mg FDC | EZ 10 mg/Atorva 20 mg FDC | Total
Number analyzed (Participants) | 117 | 18 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (12.6) | 61.6 (10.9) | 58.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 6 | 54
  Male | 69 | 12 | 81

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience 1 or More Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. The percentage of participants that reported at least 1 AE was summarized.
Time Frame: up to 54 Weeks
Population: All participants that received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | EZ 10 mg/Atorva 10 mg FDC | EZ 10 mg/Atorva 20 mg FDC
Number analyzed (Participants) | 117 | 18
Percentage of Participants | 82.9 | 88.9

2. Primary Outcome: Percentage of Participants Who Experience 1 or More Gastrointestinal-related AEs
Description: Gastrointestinal-related AEs included all preferred terms within system organ class of Gastrointestinal Disorders except Chapped Lips and Toothache.
Time Frame: up to 54 weeks
Population: All participants that received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | EZ 10 mg/Atorva 10 mg FDC | EZ 10 mg/Atorva 20 mg FDC
Number analyzed (Participants) | 117 | 18
Percentage of participants | 30.8 | 11.1

3. Primary Outcome: Percentage of Participants Who Experience 1 or More Gallbladder-related AEs
Description: Gallbladder-related AEs included Bile Duct Obstruction, Bile Duct Stone, Bile Duct Stenosis, Biliary Colic, Cholangitis, Cholecystectomy, Cholecystitis, Cholelithiasis, Gallbladder Disorder, Gallbladder Perforation, Hepatic Pain, and Hydrocholecystis.
Time Frame: up to 54 weeks
Population: All participants that received at least 1 dose of study drug and had available data for outcome.
Measure: Number; unit: Percentage of Participants
Arm/Group | EZ 10 mg/Atorva 10 mg FDC | EZ 10 mg/Atorva 20 mg FDC
Number analyzed (Participants) | 117 | 18
Percentage of Participants | 0.0 | 0.0

4. Primary Outcome: Percentage of Participants Who Experience 1 or More Allergic Reaction or Rash AEs
Description: Allergic Reaction or Rash AEs included Allergy to Arthropod Sting, Anaphylactoid Reaction, Anaphylactic Reaction, Anaphylatic Shock, Anaphylactoid Shock, Angioedema, Conjunctivitis Allergic, Contrast Media Reaction, Dermatitis, Dermatitis Allergic, Dermatitis Atopic, Dermatitis Bullous, Dermatitis Contact, Dermatitis Psoriasiform, Drug Hypersensitivity, Eczema, Eosinophila, Erythema, Eye Allergy, Face Oedema, Hypersensitivity, Mechanical Urticaria, Palmar Erythema, Periorbital Oedema, Photodermatosis, Photosensitivity Allergic reaction, Photosensitivity Reaction, Pigmentation Disorder, Pruritus, Pruritus Generalised, Rash, Rash Erythematous, Rash Follicular, Rash Generalised, Rash Maculo-Papular, Rash Papulosquamous, Rash Pruritic, Rash Pustular, Rash Vesicular, Rhinitis, Rhinitis Allergic, Rosacea, Skin Exfoliation, Skin Disorder, Skin Hyperpigmentation, Skin Lesion, Skin Mass, Skin Ulcer, Subcutaneous Nodule, Swelling Face, Systemic Lupus Erythematosus Rash, Urticaria.
Time Frame: up to 54 weeks
Population: All participants that received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | EZ 10 mg/Atorva 10 mg FDC | EZ 10 mg/Atorva 20 mg FDC
Number analyzed (Participants) | 117 | 18
Percentage of Participants | 6.8 | 22.2

5. Primary Outcome: Percentage of Participants Who Experience 1 or More Hepatitis-related AEs
Description: Hepatitis-related AEs included Cholestasis, Cytolytic Hepatitis, Hepatic Cyst, Hepatic Failure, Hepatic Lesion, Hepatic Necrosis, Hepatitis, Hepatitis Cholestatic, Hepatitis Fulminant, Hepatitis Infectious, Hepatocellular Injury, Hepatomegaly, Jaundice, Jaundice Cholestatic.
Time Frame: up to 54 weeks
Population: All participants that received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | EZ 10 mg/Atorva 10 mg FDC | EZ 10 mg/Atorva 20 mg FDC
Number analyzed (Participants) | 117 | 18
Percentage of Participants | 0.0 | 5.6

6. Primary Outcome: Percentage of Participants Who Experience Consecutive Elevations in Alanine Aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) ≥3 Times Upper Normal Limit (ULN)
Description: Participants had ALT and AST levels assessed throughout the 52 week treatment period. Participants who had 2 consecutive assessments of ALT and/or AST that were 3 x ULN or greater were recorded. The ALT and AST ULNs were 40 U/L.
Time Frame: up to 52 weeks
Population: All participants that received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | EZ 10 mg/Atorva 10 mg FDC | EZ 10 mg/Atorva 20 mg FDC
Number analyzed (Participants) | 117 | 18
Percentage of Participants | 0.9 | 0.0

7. Primary Outcome: Percentage of Participants Who Experience Elevations in ALT or AST ≥5 Times ULN
Description: Participants had ALT and AST levels assessed throughout the 52 week treatment period. Participants who had assessments of ALT or AST that were 5x ULN or greater were recorded. The ALT and AST ULNs were 40 U/L.
Time Frame: up to 52 weeks
Population: All participants that received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | EZ 10 mg/Atorva 10 mg FDC | EZ 10 mg/Atorva 20 mg FDC
Number analyzed (Participants) | 117 | 18
Percentage of Participants | 0.0 | 0.0

8. Primary Outcome: Percentage of Participants Who Experience Elevations in ALT or AST ≥10 Times ULN
Description: Participants had ALT and AST levels assessed throughout the 52 week treatment period. Participants who had assessments of ALT and/or AST that were 10x ULN or greater were recorded. The ALT and AST ULNs were 40 U/L.
Time Frame: up to 52 weeks
Population: All participants that received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | EZ 10 mg/Atorva 10 mg FDC | EZ 10 mg/Atorva 20 mg FDC
Number analyzed (Participants) | 117 | 18
Percentage of Participants | 0.0 | 0.0

9. Primary Outcome: Percentage of Participants With Potential Hy's Law Condition
Description: Percentage of Participants with Potential Hy's Law Condition (defined as serum ALT or serum AST elevations >3xULN, with serum alkaline phosphatase <2xULN and total bilirubin (TBL) ≥2xULN) was summarized. The ALT and AST ULNs were 40 U/L. The ULN for alkaline phosphatase was 359 IU/L and the ULN for total bilirubin was 1.2 mg/dL.
Time Frame: up to 52 weeks
Population: All participants that received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | EZ 10 mg/Atorva 10 mg FDC | EZ 10 mg/Atorva 20 mg FDC
Number analyzed (Participants) | 117 | 18
Percentage of Participants | 0.0 | 0.0

10. Primary Outcome: Percentage of Participants Who Experience Elevations in Creatine Kinase (CK) ≥10 Times ULN
Description: Participants had creatine phosphokinase (CK) levels assessed throughout the 12 week treatment period. Participants who had any CK level that was ≥10 x ULN were recorded. The CK ULNs for males and females were 287 IU/L and 163 IU/L, respectively.
Time Frame: up to 52 weeks
Population: All participants that received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | EZ 10 mg/Atorva 10 mg FDC | EZ 10 mg/Atorva 20 mg FDC
Number analyzed (Participants) | 117 | 18
Percentage of Participants | 0.0 | 0.0

11. Primary Outcome: Percentage of Participants Who Experience Elevations in Creatine Kinase (CK) ≥10 Times ULN With Muscle Symptoms
Description: Participants had CK levels assessed throughout the 52 week treatment period. Participants who had any CK level that was ≥10 x ULN and had associated muscle symptoms present within +/- 7 days were recorded. The CK ULNs for males and females were 287 IU/L and 163 IU/L, respectively.
Time Frame: up to 52 weeks
Population: All participants that received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | EZ 10 mg/Atorva 10 mg FDC | EZ 10 mg/Atorva 20 mg FDC
Number analyzed (Participants) | 117 | 18
Percentage of Participants | 0.0 | 0.0

12. Primary Outcome: Percentage of Participants Who Experience Elevations in Creatine Kinase (CK) ≥10 Times ULN and Drug-Related Muscle Symptoms
Description: Participants had CK levels assessed throughout the 52 week treatment period. Participants who had any CK level that was ≥10 x ULN and had associated muscle symptoms present within +/- 7 days that were reported as at least possibly-related to study drug were recorded. The CK ULNs for males and females were 287 IU/L and 163 IU/L, respectively.
Time Frame: up to 52 weeks
Population: All participants that received at least 1 dose of study drug and had available data for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | EZ 10 mg/Atorva 10 mg FDC | EZ 10 mg/Atorva 20 mg FDC
Number analyzed (Participants) | 117 | 18
Percentage of Participants | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Description: Population included all participants that received at least 1 dose of study drug.
Groups:
- EZ10/AT10: One ezetimibe (EZ) 10 mg/atorvastatin (Atorva) 10 mg fixed-dose combination (FDC) tablet orally with food once daily for 52 weeks.
- EZ10/AT20: One EZ 10 mg/Atorva 20 mg fixed -dose combination (FDC) tablet orally with food once daily for 52 weeks.
Arm/Group | EZ10/AT10 | EZ10/AT20
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/18
Serious Adverse Events (participants affected / at risk) | 7/117 | 2/18
Other Adverse Events (participants affected / at risk) | 77/117 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EZ10/AT10 (N=117) | EZ10/AT20 (N=18)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Progressive supranuclear palsy (Nervous system disorders) | 1 (1) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EZ10/AT10 (N=117) | EZ10/AT20 (N=18)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Scintillating scotoma (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 6 (6) | 0 (0)
Oral hyperaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 50 (75) | 7 (13)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 6 (6) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Electrocardiogram ST-T segment depression (Investigations) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 11 (11) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 6 (10) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Sciatica (Nervous system disorders) | 3 (3) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.